CLINICAL TRIAL: NCT01225198
Title: New Vitamin/Mineral Supplement for Children and Adults With Autism - National Study
Brief Title: Vitamin/Mineral Supplement for Children and Adults With Autism
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Arizona State University (Other)
Collaborators: Autism Research Institute (Unknown); Legacy Foundation (Unknown)
Responsible Party: James B. Adams, Arizona State University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AutismVitaminStudy2008
Record Dates: First submitted 2010-09-14; First posted 2010-10-20 (Estimated); Last update posted 2010-10-20 (Estimated); Status verified 2010-10

CONDITIONS: Autism
Keywords: Vitamins; Minerals
MeSH Terms: conditions — Autistic Disorder | interventions — Geritol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo Group (Placebo Comparator): Liquid placebo with identical packaging and flavoring to the real supplement.
  Interventions: Other: Liquid Placebo
- Vitamin/Mineral Supplement Group (Experimental): Multi-vitamin/mineral supplement designed for this study for children and adults with autism spectrum disorders.
  Interventions: Dietary Supplement: Multi-Vitamin/Mineral Supplement

INTERVENTIONS:
Dietary Supplement: Multi-Vitamin/Mineral Supplement — A broad-spectrum vitamin/mineral supplement designed for children and adults with autism
  Arms: Vitamin/Mineral Supplement Group
Other: Liquid Placebo — The placebo was formulated to look and taste like the intervention supplement. A small amount of beta-carotene was used for coloring. Natural cherry, citric acid, and a proprietary blend of natural flavors were used for flavoring to create a vitamin-like after-taste. Sucralose was used as a sweetener and the same preservatives were included (potassium sorbate, sodium benzoate).
  Arms: Placebo Group

SUMMARY:
The investigators hypothesis is that a new, revised formulation of a vitamin/mineral supplement will result in:

1. improvement of nutritional status in some children/adults with autism, and
2. reduction of some of the symptoms of autism in some children

DETAILED DESCRIPTION:
The major goal of this study is to determine the effect of this vitamin/mineral supplement on levels of vitamins, minerals, neurotransmitters, and biomarkers for nutritional deficiencies. The study design is a randomized, double-blind, placebo-controlled. Blood and urine measurements will be measured at the beginning of the study in children with autism and typical children. Then, the children with autism will be given the supplement or placebo for 12 weeks, and then their blood and urine will be re-measured.

ELIGIBILITY:
Inclusion Criteria:

1. age 3-60 years old;
2. Autism Group: diagnosis of autism, pervasive developmental disorder/not otherwise specified (PDD/NOS), or Asperger's by a psychiatrist or similar professional
3. Control Group: in good mental and physical health, and no siblings with autism spectrum disorders, and no evidence of Attention Deficit Disorder by parent report

Exclusion Criteria:

1. Usage of a vitamin/mineral supplement in the last 2 months
2. Current use of any chelation treatment

Ages: 3 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 143 (Actual)
Dates: Start 2008-05; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Oxidative Stress | Beginning of study (day 0)
  Level of Plasma Nitrotyrosine
Oxidative Stress | End of Study (after 12 weeks of treatment)
  Level of plasma nitrotyrosine

SECONDARY OUTCOMES:
Parent Global Impressions - Revised | End of study (12 weeks)
  The Average Change of the Parent Global Impressions (PGI-R) assessment tool.

CONTACTS AND LOCATIONS:
Overall Officials: James B. Adams, PhD, Principal Investigator — Arizona State University
Locations (1):
- Arizona State University, Tempe, Arizona, United States

REFERENCES:
- [Derived] Adams JB, Audhya T, McDonough-Means S, Rubin RA, Quig D, Geis E, Gehn E, Loresto M, Mitchell J, Atwood S, Barnhouse S, Lee W. Effect of a vitamin/mineral supplement on children and adults with autism. BMC Pediatr. 2011 Dec 12;11:111. doi: 10.1186/1471-2431-11-111. PMID 22151477
- See also: Arizona State University Autism/Asperger's Research Program — http://autism.asu.edu